CLINICAL TRIAL: NCT01537198
Title: Post-Marketing Surveillance of Synagis in Korean Pediatric Patients Under the "New Drug Re-Examination"
Brief Title: Surveillance of Synagis in Korean Pediatric Patients
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-203
Record Dates: First submitted 2011-12-15; First posted 2012-02-23 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-06

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: Postmarketing Drug Surveillance
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Participants at High Risk of RSV: Pediatric participants at high risk of respiratory syncytial virus (RSV) in need of the prevention of serious lower respiratory tract disease caused by RSV were prescribed Synagis prophylaxis in usual practice according to the approved Korean product label. The decision to prescribe or not to prescribe Synagis was taken prior to a participant's enrollment in the study.

SUMMARY:
Approximately 600 pediatric patients prescribed palivizumab (Synagis) prophylaxis in usual practice according to the approved Korean product label will be registered into this observational study. Baseline data will be obtained at enrollment including demographics, gestational age, birth weight and underlying diseases and complications especially in regard to respiratory disease and cardiovascular disease. At routine visits for Synagis administration, which will occur according to usual medical practice, information on Synagis prophylaxis, concomitant medication, and adverse events will be collected for up to 30 days after the last administration of Synagis.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients at high risk of RSV disease, who need the prevention of serious lower respiratory tract disease caused by RSV, and meet any of the following criteria:

  * Preterm newborn infants or infants born at 35 weeks of gestation or less, and less than 6 months of age at the onset of RSV season (RSV season defined as Oct. 1 to the following Mar. 31).
  * Newborn infants, infants, or children under 2 years of age and requiring treatment for bronchopulmonary dysplasia (BPD) within the last 6 months preceding RSV season (RSV season defined as Oct. 1 to the following Mar. 31).
  * Newborn infants, infants, or children under 2 years of age with hemodynamically significant congenital heart disease (CHD).
* Obtained authorization form to use personal and/or health data from legal representative prior to the entry into the study.

Exclusion Criteria:

* Contraindications according to the approved label.

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: General hospital
Sampling Method: Probability Sample
Enrollment: 618 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SoRa Lee, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/index.cfm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 618 participants were enrolled; 1 participant was a duplicate enrollment and the duplicate data was excluded from the analysis.
Period: Overall Study
Arm/Group | Pediatric Participants at High Risk of RSV
Started | 617
Completed | 463
Not Completed | 154
Not completed — RSV infection | 2
Not completed — Adverse Event | 4
Not completed — No Further Visits to the Clinic | 37
Not completed — Other | 111

BASELINE CHARACTERISTICS:
Groups:
- Pediatric Participants at High Risk of RSV: Pediatric participants at high risk of RSV in need of the prevention of serious lower respiratory tract disease caused by RSV were prescribed Synagis prophylaxis in usual practice according to the approved Korean product label. The decision to prescribe or not to prescribe Synagis was taken prior to a participant's enrollment in the study.
Arm/Group | Pediatric Participants at High Risk of RSV
Number analyzed (Participants) | 617
Age, Continuous [Mean (Standard Deviation); unit: months] | 3.38 (3.39)
Age, Customized [Number; unit: participants]
  Newborn infants (0 to 27 days) | 166
  Infants and toddlers (28 days to 23 months) | 451
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281
  Male | 336

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs), Serious AEs (SAEs), and Adverse Drug Reactions (ADRs)
Description: An AE was defined as any untoward medical occurrence that did not necessarily have a causal relationship with treatment. An SAE was an event that resulted in death, was life-threatening, required or prolonged hospitalization, resulted in congenital anomaly or persistent or significant disability, important medical event requiring medical or surgical intervention to prevent serious outcome, or a spontaneous or elective abortion. AEs considered to be related to Synagis were classified as ADRs. The causality of ADRs were assessed by the investigator as 'Probable,' 'Possible' and 'others (unknown). 'Unexpected' AEs are those that are unlabeled.
Time Frame: From the time of informed consent until 30 days after the final administration of Synagis, an expected average of 6 months from the start of Synagis
Measure: Number; unit: participants
Arm/Group | Pediatric Participants at High Risk of RSV
Number analyzed (Participants) | 617
participants
  Any AE | 126
  Any ADR | 3
  Any SAE | 46
  Any serious ADR | 3
  Any unexpected AE | 67
  Any unexpected ADR | 0

ADVERSE EVENTS:
Time Frame: From the time of informed consent until 30 days after the final administration of Synagis, an expected average of 6 months from the start of Synagis
Arm/Group | Pediatric Participants at High Risk of RSV
Serious Adverse Events (participants affected / at risk) | 46/617
Other Adverse Events (participants affected / at risk) | 32/617
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric Participants at High Risk of RSV (N=617)
Respiratory syncytial virus infection (Infections and infestations) | 11
Bronchiolitis (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 4
Rhinovirus infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Pneumonia adenoviral (Infections and infestations) | 1
Adenovirus infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
H1N1 influenza (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Pyrexia (General disorders) | 4
Condition aggravated (General disorders) | 3
Death (General disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Clonic convulsion (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Retinopathy of prematurity (Eye disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Cyanosis (Cardiac disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Feeding disorder neonatal (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric Participants at High Risk of RSV (N=617)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.